CLINICAL TRIAL: NCT04942223
Title: Guided Bone Regeneration With Custom Made Meshes in the Dental Rehabilitation of Three Dimensional and Extended Defect of the Jaws.
Brief Title: Guided Bone Regeneration With Custom Made Meshes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Giuseppe Lizio, research assistant, University of Bologna
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 121/2013
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: The Presence of Horizontal and Vertical Alveolar Defects in Both Jaws, Inadequate for the Placement of at Least Two Fixtures, Even ≤6 mm Long Ones
Keywords: virtual planning, GBR, titanium meshes.

STUDY DESIGN:
Intervention Model Description: prospective pilot cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects undergoing virtually planned GBR for extended and complex alveolar defects. (Other): Subjects undergoing virtually planned GBR for extended and complex alveolar defects.
  The subjects were selected from the population of patients referring to the Oral & Maxillofacial Surgery Unit of S.Orsola-Malpighi University Hospital for oral function rehabilitation. Eligibility criteria were: the presence of horizontal and vertical alveolar defects in both jaws, inadequate for the placement of at least two fixtures, even ≤6 mm long ones; ≥ 18 years; informed consent signed.
  Interventions: Device: guided bone regeneration

INTERVENTIONS:
Device: guided bone regeneration — After local anesthesia, the surgery started with a mid-crestal incision with vertical releasing cuts followed by the full-thickness buccal and lingual/palatal flaps raising to expose the bone defect completely. The flaps were coronally extended to assure a complete closure with a passive suture above the titanium. Subsequently, an intra-oral mandibular ramus bone cortical block was harvested in the molar zone. The bone block was milled and mixed with freeze-dried. The particulate graft was put to fill the deficit above the mesh until its perfect stability and unity with the defect's borders. Two or three titanium mini-screws were used to stabilize the device , and the flaps were carefully sutured. Ceftriaxone was administered intravenously at a loading dose of 2 g; together with a non-steroidal analgesic, it was continued at two g/die per os beginning the day after surgery and continuing for six days.
  Other Names: bone reconstruction

SUMMARY:
Twenty patients underwent a guided bone regenerative procedure with the application of a virtually projected customized mesh as containment and stabilizer of particulate bone graft. The entity of bone volume reconstructed after healing were digitally analysed on radiological imaging and expressed in volumetric data and in percentage of what planned before the operation. This datum was correlated with predictors variables potentially affecting the final results. As secondary outcome the implant results after the prosthetic loading was evaluated in terms of survival, success and complication.

DETAILED DESCRIPTION:
The implant-borne rehabilitation of three-dimensional and extended alveolar defects is not simple in any case: anatomic and prosthetic demands often require bone reconstructive procedures. Up to date, we can entirely virtually simulate our treatment .The design and printing of a customized mesh mimicking the ideal reconstruction eliminate the intra-operative handling and trimming, with reduced surgical timings and minimal stress for the soft tissues.

The aim is to verify if virtual planning with a customized scaffold could improve the predictability of a complex bone reconstruction in terms of bone reconstruction and implant results.

Twenty patients underwent a guided bone regenerative procedure with the application of a virtually projected customized mesh as containment and stabilizer of particulate bone graft. The entity of bone volume reconstructed after healing were digitally analysed on radiological imaging and expressed in volumetric data and in percentage of what planned before the operation. This datum was correlated with predictors variables potentially affecting the final result: six months at least after surgery, a new cone-beam CT was taken;the pre-and postoperative CT datasets were converted into three-dimensional models and digitally aligned; the reconstructed bone volumes (RBV) were calculated according to the planned bone volumes (PBVs), outlining the areas under the mesh. These values were correlated with complications, atrophies' location and the entity of virtually planned bone volume. As secondary outcome the implant results after the prosthetic loading was evaluated in terms of survival, success and complication.

ELIGIBILITY:
Inclusion Criteria:

* The presence of horizontal and vertical alveolar defects in both jaws, inadequate for the placement of at least two fixtures, even ≤6 mm long ones;
* ≥ 18 years;
* informed consent signed.

Exclusion Criteria:

* acute or chronic infections in the head and neck;
* smoking >10 cigarettes per day;
* uncontrolled diabetes (glycated hemoglobin level > 7 mg/dL);
* a history of radiation therapy in the head or neck region;
* current antitumor chemotherapy;
* liver, blood, or kidney disease;
* immunosuppression;
* everyday corticosteroid use;
* pregnancy;
* inflammatory and autoimmune disease of the oral cavity;
* poor oral hygiene and motivation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Bone regeneration volumes | 6 months after surgery
  The bone reconstruction was calculated comparing the pre-operative and postoperative volumes. The Reconstructed Bone Volume (RBV) derived by subtracting the Lacking Bone Volume (LBV) values from Planned Bone Volume (PBV) ones. The pre-and postoperative CT datasets were converted into 3D models using Amira imaging software, version 5.3.3. The segmentation regarded almost the entire jaw structure to have at least six precise anatomical points of matching for the superimposition. After that, the pre and postoperative models were digitally aligned with Geomagic Studio 12 software. After the alignment was verified at a minimum range of tolerance of error level of ±0.37 mm in the areas no involved by the surgery, the measurements were performed. In every single slice, the space between the mesh profile and the basal bone was virtually selected and rendered to obtain the PBV; the area representative for the empty space according to the gray-scale of pixels was rendered for the LBV.

SECONDARY OUTCOMES:
Implant survival. | 1 year after implant loading at least.
  The number of implants in function at the end of follow-up was recorded
Complication rate | through study completion, an average of 2 years.
  The number of complications (peri-implantitis, infections, prosthetic fractures, soft tissue problems) was recorded and expressed in numerical data.
Implant success | 1 year after implant loading at least.
  The implant succes was calculated in respect to the bone resorption around each implant, radiographically assessed: with a dedicated software, the distance between the implant shoulder and the higher point of bone-implant contact was measured mesially and distally, attributing a mean value to each implant. These measures, expressed in millimeters, were recorded and reported as numerical data.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe lizio, DDS, Principal Investigator — University of Bologna (Italy) UNIBO